CLINICAL TRIAL: NCT03053661
Title: Immune Response Evaluation to Curative Conventional Therapy of Stage III/IV Head and Neck Squamous Cell Carcinoma Patients
Brief Title: Immune Response Evaluation to Curative Conventional Therapy
Acronym: IRECT-01
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Simon Laban, MD, Head & Neck Cancer Lead, Interdisciplinary Oncologic Outpatient Unit, University of Ulm
Other Study IDs: IRECT-01
Record Dates: First submitted 2017-02-12; First posted 2017-02-15 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Squamous Cell Carcinoma; cancer-specific immunity; cancer immunology; cancer-testis antigens; human papilloma virus; immune modulatory cells
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, peripheral blood mononuclear cells, tumor tissue (fresh frozen), formalin fixed paraffin embedded tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- primary surgery + adj. C)RT: treatment naive patients to be treated by conventional primary surgery followed by adjuvant (chemo-)radiotherapy with curative intent
- primary chemoradiation: treatment naive patients to be treated by conventional primary chemoradiotherapy with curative intent

SUMMARY:
The IRECT trial is a non-interventional, prospective clinical trial using modern immune monitoring techniques over the course of the standard of care for HNSCC. The dynamics of host/tumor immune interactions during the conventional standard treatment will be analyzed to find the most promising target antigen and to develop a strategy how and when specific immunotherapy should be added to the current treatment schedule.

The results from this trial will help to understand how state of the art treatment can be complemented using cancer-testis antigen specific vaccines and immune-modulating drugs to improve the outcome of head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed patients with stage III-IVa/b head and neck squamous cell carcinoma
* fit for treatment with curative intent
* conventional primary treatment
* primary surgical treatment
* primary radiotherapeutic treatment
* informed consent
* >18 years of age
* sufficient contraception

Exclusion Criteria:

* distant metastasis at baseline
* severe concomitant disease compromising curative treatment
* previously diagnosed other malignant diseases
* active immunosuppressive therapy
* known immune defect
* pregnancy
* anemia requiring treatment at study entry (<9g/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stage III-IVa/b treatment-naive head and neck squamous cell carcinoma patients
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-08; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
prevalence of spontaneous tumor-specific immunity at baseline | baseline
dynamics of tumor-specific immunity and immune modulatory cells during conventional treatment | 7-12 weeks (treatment phase)
dynamics of tumor-specific immunity and immune modulatory cells during follow up | 12 months after end of treatment

SECONDARY OUTCOMES:
overall survival at 3 years | baseline - 3 years
progression free survival at 3 years | baseline - 3 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Witzleben A, Fehn A, Grages A, Ezic J, Jeske SS, Puntigam LK, Brunner C, Kraus JM, Kestler HA, Doescher J, Brand M, Theodoraki MN, Ottensmeier CH, Hoffmann TK, Schuler PJ, Laban S. Prospective longitudinal study of immune checkpoint molecule (ICM) expression in immune cell subsets during curative conventional therapy of head and neck squamous cell carcinoma (HNSCC). Int J Cancer. 2021 Apr 15;148(8):2023-2035. doi: 10.1002/ijc.33446. Epub 2020 Dec 30. PMID 33336372